CLINICAL TRIAL: NCT03020134
Title: Phase I Study of Pharmacokinetics and Safety of Ravidasvir in Combination With Ritonavir-boosted Danoprevir in Single and Multiple Doses in Healthy Participants
Brief Title: Pharmacokinetics and Safety of Ravidasvir and Danoprevir/r in Healthy Volunteers China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASC162002
Record Dates: First submitted 2017-01-05; First posted 2017-01-13 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: pharmacokinetics; Danoprevir/r; Ravidasvir
MeSH Terms: interventions — ravidasvir; danoprevir; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PKGroup(Ravidasvir/Danoprevir/Ritonavir) (Experimental): Ravidasvir + Danoprevir/ Ritonavir
  Interventions: Drug: Ravidasvir; Drug: Danoprevir; Drug: Ritonavir
- Placebo Group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ravidasvir — Ravidasvir tablet administered orally 200mg QD on day 1, 13 - 23
  Other Names: ASC16(RDV)
  Arms: PKGroup(Ravidasvir/Danoprevir/Ritonavir)
Drug: Danoprevir — Danoprevir tablet administered orally 100mg QD on day 7 and 13, 100mg BID on day 14-22, 100mg QD on day 23
  Other Names: ASC08 (DNV)
  Arms: PKGroup(Ravidasvir/Danoprevir/Ritonavir)
Drug: Ritonavir — Ritonavir tablet administered orally 100mg QD on day 7 and 13, 100mg BID on day 14-22, 100mg QD on day 23
  Other Names: RTV
  Arms: PKGroup(Ravidasvir/Danoprevir/Ritonavir)
Drug: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetics and safety of Ravidasvir in Combination with Ritonavir-boosted Danoprevir in Single and Multiple doses in Healthy Participants

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Overall health situation is good according to disease history, physical exam, physical symptoms, laboratory tests and 12 lead ECG.
* If female, surgically sterilized or willingness to use reliable method of birth control during the study and for 30 days after the last dose of study medication.
* If male, surgically sterilized or willingness to use reliable method of birth control during the study and for 30 days after the last dose of study medication.
* If female, negative pregnancy test during the screening period.
* Others as specified in the detailed protocol

Exclusion Criteria:

* History or presence of cardiovascular disease, respiratory disease, endocrine and metabolic system disease, urinary system, digestive system, hematological system diseases, nervous system or Psychiatric diseases, and acute or chronic infectious disease and malignant tumor.
* Positive test in any of the HAV-IgM,HBsAg, HCV Ab, HIV Ab, Syphilis Ab
* History of gastrointestinal surgery, trunk vagotomy, intestinal excision or any other surgeries that could disturb gastrointestinal motility and PH absorption.
* Female during pregnancy, breastfeeding, period and unwilling to take reliable birth control method.
* Others as specified in the detailed protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2016-08-22 (Actual); Study Completion 2016-08-22 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 40 days

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum plasma concentration at steady-state (Css,max) | Up to 24 weeks
Pharmacokinetics: Total area under the concentration-time curve form time 0 to 12 hours post-dose at steady-state | Up to 24 days

CONTACTS AND LOCATIONS:
Overall Officials: Huoling Tang, PhD, Study Director — Ascletis Pharmaceuticals Co., Ltd.

IPD SHARING:
Plan to Share IPD: No